CLINICAL TRIAL: NCT04195867
Title: Generation of Biological Samples Positive to Salmeterol for Anti-Doping Control
Acronym: SALM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IMIMFTCL/SALM
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Healthy Volunteers
Keywords: Salmeterol; Anti-doping control; Athletic performance
MeSH Terms: interventions — Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Salmeterol (Experimental): Subjects receive a 3-day treatment and collect urine from 2 days before first administration to 24 hours post-administration.
  Interventions: Drug: Salmeterol Xinafoate

INTERVENTIONS:
Drug: Salmeterol Xinafoate — Subjects receive a daily inhaled dose of 200 μg (4 inhalations of 50 μg each).

SUMMARY:
Background:

In terms of doping, there is controversy regarding the beneficial effects of β2-agonists like salmeterol on physical performance. Some studies show improvement with salmeterol administered orally, especially related to pulmonary function and muscle contractibility, while other works do not show such ergogenic effects of salmeterol by inhalation.

Supratherapeutic use of salmeterol is prohibited by the World Anti-Doping Agency, but a maximum allowed urine concentration has not been determined.

Urine concentrations of salmeterol are very low when administered at therapeutic doses, often below the lower limit of quantification. Some studies show that urine concentrations of α-hydroxy-salmeterol (the principal salmeterol metabolite) may be higher than those of the original drug. Thus, α-hydroxy-salmeterol might be a more suitable biomarker for detecting fraudulent use of this drug.

Hypothesis:

Inhaled administration of salmeterol in healthy subjects allows obtaining positive urine samples that will be used to identify analytical strategies for doping detection. Salmeterol concentrations and its metabolites (α-hydroxy-salmeterol and others) can be measured in urine.

Objectives:

Primary objective: To generate urine samples positive to salmeterol in order to be analyzed as control samples by anti-doping laboratories.

Secondary objectives: To identify salmeterol metabolites (α-hydroxy-salmeterol and others) in urine.

Methods:

Phase I, open, non-randomized, uncontrolled clinical trial, with a treatment condition (salmeterol) administered daily by inhalation to 6 subjects during 3 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers aged between 18 and 45 years.
* Able to understand and accept the trial procedures and able to sign an informed consent.
* History and physical examination that demonstrate not presenting organic or psychiatric disorders.
* ECG, blood and urine tests performed at screening should be within normal limits. Minor or punctual variations of these limits of normality are admitted if, in the opinion of the Principal Investigator, they have no clinical significance, do not pose a risk to the subject and do not interfere with the evaluation of the product in study. These variations and their non-relevance will be justified in writing specifically.
* Body mass index (weight/size^2) between 19 and 26 kg/m2, and weight between 50 and 90 kg. Subjects with BMI >27 kg/m2 may be included at the discretion of the Principal Investigator.

Exclusion Criteria:

* Failure to meet the inclusion criteria.
* History of allergy, idiosyncrasy, hypersensitivity or adverse reactions to the active substance or any of the excipients. History of serious adverse reactions to other medications.
* Subjects with contraindications to treatment with the study drug (according to Summary of Product Characteristics).
* Background or clinical evidence of psychiatric disorders, alcoholism, regular consumption of psychoactive drugs, drug abuse or addiction to other substances (except for nicotine). Smokers of more than 5 cigarettes/day will be excluded.
* Having participated in another clinical trial with medication in the three months prior to the start of the study.
* Having donated blood during the month prior to the start of the study.
* Having suffered an organic disease or major surgery in the three months prior to the start of the study.
* Background or clinical evidence of cardiovascular, respiratory (especially asthma or Chronic Obstructive Pulmonary Disease), renal, hepatic, endocrine, gastrointestinal, hematological, neurological, dermatological or other acute or chronic diseases that, in the opinion of the Principal Investigator or the collaborators designated by him, may pose a risk to the subjects, may interfere with the objectives of the study or may alter the pharmacokinetics of the drug.
* Have taken medication regularly in the month prior to the study sessions, with the exception of vitamins, herbal remedies or dietary supplements that, in the opinion of the Principal Investigator or the collaborators designated by him, do not pose a risk to the subjects and do not interfere with the objectives of the study. Treatment with single doses of symptomatic medication in the week prior to the study sessions will not be exclusive if it is assumed that medication has been completely eliminated on the day of the experimental session.
* Consumption of more than 15 g of alcohol per day.
* Consumers of more than 3 coffees, teas, cola drinks and/or other stimulant drinks (xanthines) per day in the month prior to the start of the study.
* Being unable to understand the nature of the trial and the procedures requested to follow.
* Positive serology for hepatitis B, C or HIV.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Changes in urine concentration of salmeterol | From 0 hours after first administration to 48 hours after third administration
  Variation of the concentration of salmeterol in urine

SECONDARY OUTCOMES:
Changes in urine concentration of α-hydroxy-salmeterol | From 0 hours after first administration to 48 hours after third administration
  Variation of the concentration of α-hydroxy-salmeterol in urine
Changes in urine concentrations of other salmeterol metabolites | From 0 hours after first administration to 48 hours after third administration
  Variation of the concentration of other salmeterol metabolites in urine

CONTACTS AND LOCATIONS:
Overall Officials: Julián A Mateus Rodríguez, MD, Study Director — IMIM (Hospital del Mar Medical Research Institute)
Locations (1):
- IMIM (Hospital del Mar Medical Research Institute), Barcelona, Spain